CLINICAL TRIAL: NCT03617939
Title: Total Cancer Care Protocol: A Lifetime Partnership With Patients Who Have or May be at Risk of Having Cancer (ORIEN)
Brief Title: A Lifetime Partnership With Patients Who Have or May be at Risk of Having Cancer
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 15-1110.cc
Record Dates: First submitted 2018-07-03; First posted 2018-08-07 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Cancer Risk
Keywords: Tissue Repository; Blood Samples; Biological Samples; Surveys; Early Detection; Risk Assessment

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Biospeciman and Data Collection: Patients with cancer or who are at risk of having cancer who have given consent to have blood, tissue, other biological samples and their associated data (survey data, medical records data, cancer registry data, and other related data) collected and stored for the advancement of medicine.
  Interventions: Procedure: Biospeciman Collection; Other: Survey Assessments; Other: Medical Chart Reviews

INTERVENTIONS:
Procedure: Biospeciman Collection — Collection of blood, tissue, and other biological samples.
Other: Survey Assessments — Data taken from patient surveys and assessments, including quality of life.
Other: Medical Chart Reviews — Data taken directly from the patients' medical charts.

SUMMARY:
This is not a treatment study. The overall objective is to develop an improved standard of care through studying blood, tissue, biological, etc. samples, that patients have allowed researchers to procure.

DETAILED DESCRIPTION:
The Oncology Research Information Exchange Network (ORIEN) hopes to establish a unique collection of blood, tissue, other biological samples and their associated data (survey data, medical records data, cancer registry data, and other related data) from thousands of patients with cancer or at risk of having cancer. Their hope is to, over time, facilitate new clinical trials, technology, informatics solutions, and personalized medicine to each cancer patient.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age and older.
2. Diagnosed with cancer, or may be at risk for cancer.
3. Able to understand and sign the TCCP Informed Consent and Research Authorization form directly or through a legally authorized representative (LAR).

Non-English speaking subjects will also be invited to participate in the TCCP study, in accordance with COMIRB's short-form consent use.

Exclusion Criteria:

1. Members of vulnerable populations including neonates (birth to 30 days), children (under age 18), wards of the State, prisoners or those on probation or alternate sentencing, or decisionally challenged (adults or children that are cognitively impaired, incompetent to consent, proxy consent, or consenting in life threatening situations).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All persons who are diagnosed with cancer or at risk for cancer.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2015-09-16 (Actual); Primary Completion 2035-09 (Estimated); Study Completion 2037-09 (Estimated)

PRIMARY OUTCOMES:
Improve Standard of Cancer Care | Up to 20 years
  Establish a longitudinal clinical and related data and tissue repository that will contain patient demographics via surveys and questionnaires.
Improve Standard of Cancer Care | Up to 20 years
  Establish a longitudinal clinical and related data and tissue repository that will contain medical histories via surveys and questionnaires.
Improve Standard of Cancer Care | Up to 20 years
  Establish a longitudinal clinical and related data and tissue repository that will contain cancer predisposing risk factors via surveys and questionnaires.
Improve Standard of Cancer Care | Up to 20 years
  Establish a longitudinal clinical and related data and tissue repository that will contain quality of life care via surveys and questionnaires
Improve Standard of Cancer Care | Up to 20 years
  Establish a longitudinal clinical and related data and tissue repository that will contain blood samples from consenting patients.
Improve Standard of Cancer Care | Up to 20 years
  Establish a longitudinal clinical and related data and tissue repository that will contain tissue samples from consenting patients
Improve Standard of Cancer Care | Up to 20 years
  Establish a longitudinal clinical and related data and tissue repository that will contain other biological samples from consenting patients

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Borges, MD, Principal Investigator — University of Colorado, Denver
Locations (6):
- United States (6):
  - University of Colorado Hospital, Aurora, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - UCHealth Memorial Hospital North, Colorado Springs, Colorado
  - Cherry Creek Medical Center, Denver, Colorado
  - UCHealth Poudre Valley Health System, Fort Collins, Colorado
  - Highlands Ranch Medical Center, Highlands Ranch, Colorado